CLINICAL TRIAL: NCT01340664
Title: A Randomized, Double-Blind, Placebo-Controlled, 3-Arm, Parallel-Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Canagliflozin in the Treatment of Subjects With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin
Brief Title: An Efficacy, Safety, and Tolerability Study of Canagliflozin in the Treatment of Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin Monotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017914; 28431754DIA2003 (Other: Janssen Research & Development, LLC); 2010-024256-28 (EudraCT Number)
Record Dates: First submitted 2011-04-21; First posted 2011-04-22 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Canagliflozin; Placebo; Metformin; Hemoglobin A1c; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Canagliflozin 50 mg bid (Experimental): Each patient will receive 50 mg canagliflozin twice daily for 18 weeks.
  Interventions: Drug: Canagliflozin 50 mg; Drug: Metformin
- Canagliflozin 150 mg bid (Experimental): Each patient will receive 150 mg canagliflozin twice daily for 18 weeks
  Interventions: Drug: Canagliflozin 150 mg; Drug: Metformin
- Placebo (Placebo Comparator): Each patient will receive matching placebo twice daily for 18 weeks
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: Canagliflozin 50 mg — One canagliflozin 50-mg capsule taken orally twice daily with a meal for 18 weeks
  Arms: Canagliflozin 50 mg bid
Drug: Placebo — 1 placebo capsule taken orally twice daily with a meal for 18 weeks
  Arms: Placebo
Drug: Canagliflozin 150 mg — 1 canagliflozin 150-mg capsule taken orally twice daily with a meal for 18 weeks
  Arms: Canagliflozin 150 mg bid
Drug: Metformin — The patient's stable daily dose of Metformin background therapy should be continued throughout the study.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 2 different doses of canagliflozin compared with placebo in patients with type 2 diabetes mellitus who are receiving treatment with metformin monotherapy (ie, treatment with a single drug) and have inadequate glycemic (blood sugar) control.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither the patient nor the study doctor will know the identity of assigned study drug), placebo-controlled, parallel-group,3-arm (3 treatment groups) multicenter study to determine the efficacy, safety, and tolerability of canagliflozin compared to placebo (a capsule that is identical in appearance to canagliflozin but does not contain active drug) in patients with type 2 diabetes mellitus (T2DM) who are not achieving an adequate response from current antihyperglycemic therapy with metformin to control their diabetes. Canagliflozin (a Sodium-Glucose Cotransporter 2 inhibitor) is currently under development to lower blood sugar levels in patients with T2DM. Patients will take single-blind placebo capsules orally (by mouth) for 2 weeks before randomization. Patients will be randomly assigned canagliflozin or matching placebo, orally, twice daily, with 1 capsule taken with the morning meal and 1 capsule taken with the evening meal (2 capsules per day) and concurrent with metformin, if applicable, for up to 18 weeks. The dosing time of metformin should remain the same throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of T2DM and be currently treated with metformin
* Patients in the study must have a HbA1c between >=7 and <=10.5%
* Patients must have a fasting plasma glucose (FPG) <270 mg/dL (15 mmol/L)

Exclusion Criteria:

* History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta cell transplantation, diabetes secondary to pancreatitis or pancreatectomy, or a severe hypoglycemic episode within 6 months before screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (61):
- United States (26):
  - Little Rock, Arkansas
  - National City, California
  - Spring Valley, California
  - Bradenton, Florida
  - Marianna, Florida
  - Savannah, Georgia
  - Avon, Indiana
  - Valparaiso, Indiana
  - Madisonville, Kentucky
  - Metairie, Louisiana
  - Charlotte, North Carolina
  - Columbus, Ohio
  - Mason, Ohio
  - Perrysburg, Ohio
  - Tulsa, Oklahoma
  - Yukon, Oklahoma
  - Oregon City, Oregon
  - Pittsburgh, Pennsylvania
  - East Providence, Rhode Island
  - Nashville, Tennessee
  - Houston, Texas
  - Pearland, Texas
  - San Antonio, Texas
  - Bountiful, Utah
  - Virginia Beach, Virginia
  - Milwaukee, Wisconsin
- Canada (5):
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Brampton, Ontario
  - Toronto, Ontario
  - Saskatoon, Saskatchewan
- Czechia (7):
  - Beroun
  - Olomouc
  - Ostrava
  - Pardubice
  - Písek
  - Prague
  - Znojmo
- Mexico (4):
  - Aguascalientes
  - Guadalajara, Jalisco.
  - Monterrey
  - Tampico
- Romania (6):
  - Bacau
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Galati
  - Târgu Mureş
- Russia (7):
  - Kursk
  - Moscow
  - Saint Petersburg
  - Samara
  - Saratov
  - Tyumen
  - Voronezh
- Slovakia (6):
  - Banská Bystrica
  - Bratislava
  - Košice
  - Prešov
  - Šahy
  - Trebišov

REFERENCES:
- [Derived] Qiu R, Capuano G, Meininger G. Efficacy and safety of twice-daily treatment with canagliflozin, a sodium glucose co-transporter 2 inhibitor, added on to metformin monotherapy in patients with type 2 diabetes mellitus. J Clin Transl Endocrinol. 2014 May 5;1(2):54-60. doi: 10.1016/j.jcte.2014.04.001. eCollection 2014 Jun. PMID 29159083

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus with inadequate control despite treatment with metformin. The study was conducted between 27 June 2011 and 20 April 2012 and recruited patients from 60 study centers located in 7 countries worldwide.
Pre-assignment Details: A total of 279 patients were randomly allocated to the 3 treatment arms in the study. All 279 patients received at least 1 dose of study drug and were included in the modified intent-to-treat analysis set which was used for the efficacy and safety analyses.
Groups:
- Placebo: Each patient received matching placebo twice daily for 18 weeks.
- Canagliflozin 50 mg Bid: Each patient received 50 mg canagliflozin twice daily for 18 weeks.
- Canagliflozin 150 mg Bid: Each patient received 150 mg canagliflozin twice daily for 18 weeks.
Period: Overall Study
Arm/Group | Placebo | Canagliflozin 50 mg Bid | Canagliflozin 150 mg Bid
Started | 93 | 93 | 93
Completed | 86 | 85 | 80
Not Completed | 7 | 8 | 13
Not completed — Adverse Event | 0 | 1 | 7
Not completed — Lost to Follow-up | 2 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 4 | 0
Not completed — Glycemic withdrawal criteria | 2 | 0 | 0
Not completed — Creatinine or eGFR withdrawal criteria | 0 | 1 | 2
Not completed — Other | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 50 mg Bid | Canagliflozin 150 mg Bid | Total
Number analyzed (Participants) | 93 | 93 | 93 | 279
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 79 | 69 | 75 | 223
  >=65 years | 14 | 24 | 18 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9.32) | 58.6 (8.88) | 56.7 (10.33) | 57.4 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 53 | 49 | 149
  Male | 46 | 40 | 44 | 130
Region Enroll [Number; unit: participants]
  CANADA | 17 | 11 | 12 | 40
  CZECH REPUBLIC | 2 | 4 | 6 | 12
  MEXICO | 10 | 12 | 10 | 32
  ROMANIA | 13 | 15 | 9 | 37
  RUSSIAN FEDERATION | 18 | 17 | 20 | 55
  SLOVAKIA | 10 | 9 | 11 | 30
  UNITED STATES | 23 | 25 | 25 | 73

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 18
Description: The table below shows the least-squares (LS) mean change in HbA1c from Baseline to Week 18 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 18
Population: This analysis used the modified intent-to-treat analysis set (all patients who were randomly assigned to a treatment group and received at least 1 dose of study drug). The last-observation-carried-forward method was applied when Week 18 values were missing. The table includes only patients with both baseline and post baseline values.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Canagliflozin 50 mg Bid | Canagliflozin 150 mg Bid
Number analyzed (Participants) | 92 | 90 | 91
Percent | -0.01 (0.069) | -0.45 (0.070) | -0.61 (0.069)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg Bid; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.44, 95% CI 2-sided [-0.637 to -0.251], Standard Error of Mean 0.098
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 150 mg Bid; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.60, 95% CI 2-sided [-0.792 to -0.407], Standard Error of Mean 0.098

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 18
Description: The table below shows the least-squares (LS) mean change in FPG from Baseline to Week 18 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 18
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Canagliflozin 50 mg Bid | Canagliflozin 150 mg Bid
Number analyzed (Participants) | 92 | 90 | 91
mg/dL | 8.1 (3.291) | -15.5 (3.327) | -15.9 (3.313)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg Bid; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Sqaures Mean Difference = -23.6, 95% CI 2-sided [-32.78 to -14.38], Standard Error of Mean 4.673
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 150 mg Bid; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Sqaures Mean Difference = -24.0, 95% CI [-33.18 to -14.83], Standard Error of Mean 4.661

3. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 18
Description: The table below shows the least-squares (LS) mean percent change in body weight from Baseline to Week 18 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 18
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 50 mg Bid | Canagliflozin 150 mg Bid
Number analyzed (Participants) | 92 | 90 | 91
Percent change | -0.6 (0.3) | -2.8 (0.3) | -3.2 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg Bid; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.2, 95% CI 2-sided [-3.1 to -1.3], Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 150 mg Bid; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.6, 95% CI 2-sided [-3.5 to -1.7], Standard Error of Mean 0.5

4. Secondary Outcome: Percentage of Patients With HbA1c <7% at Week 18
Description: The table below shows the percentage of patients with HbA1c <7% at Week 18 in each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the percentage.
Time Frame: Week 18
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Canagliflozin 50 mg Bid | Canagliflozin 150 mg Bid
Number analyzed (Participants) | 92 | 90 | 91
Percentage of Participants | 31.5 | 47.8 | 57.1
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg Bid; Test type: Superiority or Other; p = 0.013, Regression, Logistic; Odds Ratio (OR) = 2.43, 95% CI 2-sided [1.21 to 4.90]
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 150 mg Bid; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.38, 95% CI 2-sided [1.68 to 6.81]

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the duration of the study; each patient participated in the study for approximately 18 weeks.
Description: Only patients who had at least one of the treatment-emergent adverse events listed in the "Other (non-Serious) Adverse Event" table are included in the total number of patients with non-serious adverse Events.
Arm/Group | Placebo | Canagliflozin 50 mg Bid | Canagliflozin 150 mg Bid
Serious Adverse Events (participants affected / at risk) | 1/93 | 0/93 | 3/93
Other Adverse Events (participants affected / at risk) | 0/93 | 0/93 | 0/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=93) | Canagliflozin 50 mg Bid (N=93) | Canagliflozin 150 mg Bid (N=93)
Oroantral fistula (Gastrointestinal disorders) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. Expedited reviews will be arranged for abstracts, poster presentations, or other materials. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.